CLINICAL TRIAL: NCT06543446
Title: Comparative Effectiveness of Prophylactic ICD Versus Non-ICD Therapy in Contemporary Heart Failure Patients With a Low Risk for Arrhythmic Death
Brief Title: Comparative Effectiveness of Prophylactic ICD Versus Non-ICD Therapy
Acronym: CONTEMP-ICD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Ilan Goldenberg, Professor of Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADVARRA
Record Dates: First submitted 2024-07-25; First posted 2024-08-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Implantable cardioverter defibrillator; Sudden cardiac death; guideline directed medical therapy
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-ICD implantation (No Intervention): No-ICD implantation despite current recommendation
- ICD implantation (Active Comparator): ICD implantation based on current guidelines
  Interventions: Procedure: ICD implantation

INTERVENTIONS:
Procedure: ICD implantation — Surgical implant of ICD device
  Arms: ICD implantation

SUMMARY:
The investigators aim to compare the risk of mortality of Non-implantable carioverter defibrillator (ICD) vs. ICD management in patients with heart failure with reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
The proposed CONTEMP-ICD trial is a prospective, multicenter, open-label, randomized controlled trial; enrolling 3290 participants with HFrEF, on stable and optimal guideline-directed medical therapy (GDMT), who are eligible for a primary prevention ICD, but have a low predicted arrhythmic risk. Enrolled participants will be randomized in a 1:1 ratio to non-ICD vs. ICD treatment arms. The investigators hypothesize that, in participants with HFrEF who have a low predicted arrhythmic risk, non-ICD vs. ICD is non-inferior with respect to the primary endpoint of all-cause mortality and superior survival free of major cardiovascular (CV) events.

This study will recruit adults 18 years of age and older with heart failure. Participants will be asked to complete questionnaires. Information from medical records will be gathered including medical history, physical exam, medications, blood work results, and imaging. Visits will be at initial, three, six months, and every six months beyond six months. For those who get an ICD device an interrogation will be collected at the visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (no upper limit)
* Class I or IIa indication for a primary prevention ICD15: Ischemic or non-ischemic cardiomyopathy and NYHA Class ≥ II if most recent LVEF is ≤ 35% OR ischemic cardiomyopathy with NYHA Class I if most recent LVEF is ≤ 30%
* Most recent LVEF (%) obtained per cardiac imaging obtained at any time prior to enrollment after being stable on optimal GDMT** for at least one month
* Stable optimal GDMT at least one calendar month prior to last cardiac imaging test, prespecified as one of the following for at least 1 calendar month prior to study randomization:

receiving all 4 therapy classes (beta-blockers, ARNI/ARB/ACE, MRA and SGLT2i) OR GDMT Score ≥ 6 (per Figure 7)

• MADIT-ICD Benefit Score < 50 (per Figure 4)

Exclusion Criteria:

* Existing ICD/CRT-D
* • Planned CRT-P or CRT-D implant for any indications including Class I or IIa indication for CRT: Presence of left bundle branch block (LBBB) with QRS ≥ 120 msec OR QRS duration ≥ 150 msec regardless of QRS morphology OR decision for CRT implant by EP provider for other indications
* Acute MI within the past 3 calendar months
* Chronic renal failure requiring hemodialysis
* Coronary revascularization within the past 3 calendar months
* History of sustained VT or VF
* Known genetic cause of cardiomyopathy
* Life expectancy < 1 year
* Unable or unwilling to follow study protocol
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3290 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | through study completion, an average of 3.5 year
  Death from any cause

SECONDARY OUTCOMES:
Major adverse cardiovascular events | through study completion, an average of 3.5 years
  First occurrence of hospitalization for one of the following: stroke, myocardiac infarction, device-related complications, ICD shocks.
Healthcare utilization | through study completion, an average of 3.5 year
  Total number of the following events during following: all-cause hospital admissions, emergency department visits, planned and unplanned clinic visits. All events will be captured from electronic medical records
Quality of life, using the Kansas City Cardiomyopathy Questionnaire [KCCQ] and EuroQol-5 Dimension (EQ-5D) | One year
  Kansas City Cardiomyopathy Questionnaire [KCCQ] (the KCCQ ranges from 0 to 100, with 0 representing the worst possible health status and 100) and EuroQol-5 Dimension (EQ-5D) (Range from -0.59 to 1, with 1 representing the best possible health state and an index value of less than 0 representing the worst possible health state)
Quality of life, using the EuroQol-5 Dimension (EQ-5D) | One year
  Range from -0.59 to 1, with 1 representing the best possible health state and an index value of less than 0 representing the worst possible health state

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Goldenberg, MD, Principal Investigator — Univ of Rochester Medical Center, Clinical Cardiovascular Research Center
Locations (15):
- United States (13):
  - MaineHealth, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Corewell Health, Grand Rapids, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Rutgers, New Brunswick, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - Northwell Health, New York, New York
  - Nuvance Health Hudson Valley Cardiovascular Practice, PC, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - Intermountain Health Care, Inc., Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

REFERENCES:
- [Background] Fiuzat M, Hamo CE, Butler J, Abraham WT, DeFilippis EM, Fonarow GC, Lindenfeld J, Mentz RJ, Psotka MA, Solomon SD, Teerlink JR, Vaduganathan M, Vardeny O, McMurray JJV, O'Connor CM. Optimal Background Pharmacological Therapy for Heart Failure Patients in Clinical Trials: JACC Review Topic of the Week. J Am Coll Cardiol. 2022 Feb 8;79(5):504-510. doi: 10.1016/j.jacc.2021.11.033. PMID 35115106
- [Derived] Goldenberg I, Zareba W, Ezekowitz JA, Albert C, Alexis JD, Anderson L, Behr ER, Daubert J, Di Palo KE, Ellenbogen KA, Dzikowicz DJ, Harrington JM, Hsich E, Huang DT, Januzzi JL, Jawaid A, Kutyifa V, Lala-Trindade A, Nakonechnyi A, Onwuanyi A, Pina IL, Sandhu RK, Sears S, Sroubek J, Baykaner T, Strawderman R, Beck C, Butler J. Rationale and design of the comparative effectiveness of ICD vs non-ICD therapy in contemporary heart failure patients at a low risk for arrhythmic death (CONTEMP-ICD) trial. Am Heart J. 2026 Jan;291:162-174. doi: 10.1016/j.ahj.2025.08.020. Epub 2025 Sep 4. PMID 40914445